CLINICAL TRIAL: NCT00293189
Title: Gene-Polymorphies in the P2X7 Gene in Patients With Osteoporotic Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Collaborators: Hvidovre University Hospital (Other)
Other Study IDs: (KF) 01 272008
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2006-05-24 (Estimated); Status verified 2005-08

CONDITIONS: Hip Fracture
Keywords: hip fracture; epidemiology; genetics; p2x7
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
We are looking after gene-polymorphies in the p2x7-gene in patient with osteoporotic fractures.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture, no dementia, low energy fracture

Exclusion Criteria:

* high energy fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Steen A Schmidt, md, Study Chair — Dept of Orthopaedics, Kolding Sygehus
Locations (1):
- Dept of orthopaedics, Kolding Sygehus, Kolding, Denmark